CLINICAL TRIAL: NCT01810575
Title: A Study to Assess the Relative Efficacy and Safety of a Single Dose of Alprostadil Cream Combined With 2 Concentrations of WC3036 Compared to Vehicle in Subjects With Erectile Dysfunction
Brief Title: Efficacy & Safety of Single Dose Alprostadil Cream (2 Concentrations Enhancer) to Vehicle in Men w/Erectile Dysfunction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Re-assessment of study
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PR-13311
Record Dates: First submitted 2013-02-27; First posted 2013-03-13 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- WC3036-11F/Alprostadil in Vehicle 2.5% (Active Comparator): Treatment A
  Interventions: Drug: WC3036-11F/Alprostadil in Vehicle 2.5%
- WC3036-12F/Alprostadil in Vehicle 0.5% (Experimental): Treatment B
  Interventions: Drug: WC3036-12F/Alprostadil in Vehicle 0.5%
- WC3036-13P/Vehicle Only 0.5% (Placebo Comparator): Treatment C
  Interventions: Drug: WC3036-13P/Vehicle Only 0.5%

INTERVENTIONS:
Drug: WC3036-11F/Alprostadil in Vehicle 2.5% — 330 mcg alprostadil in 2.5% vehicle
  Other Names: 11F
  Arms: WC3036-11F/Alprostadil in Vehicle 2.5%
Drug: WC3036-12F/Alprostadil in Vehicle 0.5% — 330 mcg alprostadil in 0.5% vehicle
  Other Names: 12F
  Arms: WC3036-12F/Alprostadil in Vehicle 0.5%
Drug: WC3036-13P/Vehicle Only 0.5% — 100 mg cream vehicle 0.5%.
  Other Names: Vehicle
  Arms: WC3036-13P/Vehicle Only 0.5%

SUMMARY:
The purpose of this study is to assess the safety & efficacy of a single dose of alprostadil cream with 2 concentrations of WC3036 compared to vehicle alone in men with erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Male subject aged 40 or older of any race
* History of ED (erectile dysfunction) of at least 3 months duration defined as inability to attain & maintain an erection of the penis sufficient to permit satisfactory sexual intercourse
* Completed and signed informed consent prior to any study related procedures

Exclusion Criteria:

* History/presence any significant disease that Investigator feels will interfere with course of the study
* Anatomic deformity of penis
* History/presence alcoholism or drug abuse/dependence within past 2 years (discretion of Investigator)
* Participation in investigational study drug trial within 30 days prior to randomization

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Penile rigidity | Visit 1 / Up to 5 days ± 3 days
  ≥60% at base and tip of penis lasting for ≥ 5 minutes evaluated with RigiScan. Treatment visits will be separated by at least 2 days.
Penile rigidity | Visit 2 / Up to 9 days ± 3 days
  ≥60% at base and tip of penis lasting for ≥ 5 minutes evaluated with RigiScan. Treatment visits will be separated by at least 2 days.
Penile rigidity | Visit 3 / Up to 14 Days
  ≥60% at base and tip of penis lasting for ≥ 5 minutes evaluated with RigiScan. Treatment visits will be separated by at least 2 days.

SECONDARY OUTCOMES:
Quality of erection | Visit 1 / Up to 5 days ± 3 days
  Subject description of quality of erection using non-validated questionnaire. Treatment visits will be separated by at least 2 days.
Quality of erection | Visit 2 / Up to 9 days ± 3 days
  Subject description of quality of erection using non-validated questionnaire. Treatment visits will be separated by at least 2 days.
Quality of erection | Visit 3 / Up to 14 days
  Subject description of quality of erection using non-validated questionnaire. Treatment visits will be separated by at least 2 days.

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Sniukiene, MD, Study Director — Warner Chilcott
Locations (1):
- Warner Chilcott Investigational Study Site, Purchase, New York, United States